CLINICAL TRIAL: NCT01604915
Title: Comparison of Analgesic Effect of Dexamethasone Added to Ropivacaine and Ropivacaine Alone in Caudal Analgesia on Postoperative Pain Control in Pediatric Patients Undergoing Orchiopexy
Brief Title: Comparison of Dexamethasone Added to Ropivacaine and Ropivacaine Alone in Caudal Analgesia in Children Undergoing Orchiopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jeong-Rim LEE, Assistant Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2012-0149
Record Dates: First submitted 2012-05-18; First posted 2012-05-24 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Cryptorchidism
MeSH Terms: conditions — Cryptorchidism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group R (Placebo Comparator): Normal saline 0.02mL/Kg added to ropivacaine 0.15% 1.5ml/kg was administered.
  Interventions: Procedure: Caudal block
- Group DR (Experimental): Dexamethasone 0.1mg/kg added to ropivacaine 0.15% 1.5ml/kg to Group DR.
  Interventions: Procedure: Caudal block

INTERVENTIONS:
Procedure: Caudal block — After inhalation induction of general anesthesia, caudal block was applied. Patients were randomly assigned in two groups. Normal saline 0.02mL/Kg added to ropivacaine 0.15% 1.5ml/kg was administered to Group R.
  Arms: Group R
Procedure: Caudal block — After inhalation induction of general anesthesia, caudal block was applied. Patients were randomly assigned in two groups. Dexamethasone 0.1mg/kg added to ropivacaine 0.15% 1.5ml/kg to Group DR.
  Arms: Group DR

SUMMARY:
Single shot caudal epidural block is one of the most widespread technique for pediatric pain management after infraumbilical surgical procedures.

However, in a significant proportion of patients, despite good initial analgesia from a caudal block with local anesthetic, pain develops after the block resolves.

In order to decrease postoperative analgesic requirements after caudal block, various drugs such as opioids, ketamine, clonidine, or dexmedetomidine to local anesthetics has been investigated. However, their use has been limited by adverse effects in children.

Recently, many study suggested that epidurally administered dexamethasone could reduce the incidence and severity of postoperative pain in adults. But there is no study concerning the use of dexamethasone, as an adjuvant agent for the caudal epidural block in children.

The investigators performed prospective randomized double-blind study to examine the analgesic effect of dexamethasone added to ropivacaine and ropivacaine alone in caudal analgesia on postoperative pain control in pediatric patients undergoing orchiopexy.

80 children (aged 0.5-5 yr) undergoing day-case orchiopexy were included in this prospective, randomized, double-blinded study. After inhalation induction of general anesthesia, caudal block was applied. Patients were randomly assigned in two groups. Normal saline 0.02mL/Kg added to ropivacaine 0.15% 1.5ml/kg was administered to Group R , dexamethasone 0.1mg/kg added to ropivacaine 0.15% 1.5ml/kg to Group DR. Postoperative pain was recorded at 30min and 1,2,3 h by using Hospital of Eastern Ontario Pain Scale (CHEOPS, 0-10) and Faces Legs Activity Cry Consolability tool (FLACC, 0-10). Participants will be followed for the duration of hospital stay, an expected average of 3 hours.

After discharge, rescue analgesic consumption, pain scores, and adverse effects were evaluated for 24h.

The time to first supplemental oral analgesic medication demand was defined as the time from the end of surgery to the first registration of a VAS ( 0-10) ≥ 5 by parent's observation. Twenty-four hours after surgery, reports of delayed side effects and demands for rescue analgesics from the child were gathered from parents via a telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I-II
* Children aged 6 months to 5 years
* Undergoing day-case unilateral orchiopexy

Exclusion Criteria:

* Hypersensitivity to any local anesthetics
* Bleeding diathesis
* Infections at puncture sites
* Preexisting neurological disease
* Diabetes mellitus

Ages: 6 Months to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Time to first analgesic rescue medication | from the end of surgery to the first registration of a VAS(0-10) ≥ 5 by parent's observation
  The time to first supplemental oral analgesic medication demand was defined as the time from the end of surgery to the first registration of a VAS ( 0-10) ≥ 5 by parent's observation. Twenty-four hours after surgery, reports of delayed side effects and demands for rescue analgesics from the child were gathered from parents via a telephone interview.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Khafagy HF, Refaat AI, El-Sabae HH, Youssif MA. Efficacy of epidural dexamethasone versus fentanyl on postoperative analgesia. J Anesth. 2010 Aug;24(4):531-6. doi: 10.1007/s00540-010-0949-7. Epub 2010 May 14. PMID 20467878
- [Derived] Kim EM, Lee JR, Koo BN, Im YJ, Oh HJ, Lee JH. Analgesic efficacy of caudal dexamethasone combined with ropivacaine in children undergoing orchiopexy. Br J Anaesth. 2014 May;112(5):885-91. doi: 10.1093/bja/aet484. Epub 2014 Feb 2. PMID 24491414